CLINICAL TRIAL: NCT06558461
Title: Evaluating the Efficacy of Nebulised 3% Hypertonic Saline for Acute Bronchiolitis in Infants: A Study at Can Tho Children's Hospital, 2022-2024
Brief Title: Nebulised 3% Hypertonic Saline in Infants With Acute Bronchiolitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 173
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Acute Bronchiolitis
Keywords: Bronchiolitis; 3% hypertonic saline
MeSH Terms: conditions — Bronchiolitis | interventions — Sodium Chloride; Standard of Care

STUDY DESIGN:
Intervention Model Description: A randomized controlled open-label parallel-arm clinical trial, with allocation 1:1, was conducted to investigate whether nebulizing 3% hypertonic saline will improve clinical symptoms and reduce the length of hospital stay in bronchiolitis compared with the control group.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 3% hypertonic saline (Experimental): Children will receive standard medical care coordinating with nebulizing 3% hypertonic saline in the treatment of bronchiolitis. They received 4ml of 3% Sodium chloride, nebulized three times daily until discharge.
  Interventions: Drug: 3% Sodium Chloride
- Control (Active Comparator): Children will only receive standard medical care.
  Interventions: Other: Standard care

INTERVENTIONS:
Drug: 3% Sodium Chloride — 4ml nebulized three times daily
  Arms: 3% hypertonic saline
Other: Standard care — Standard care
  Arms: Control

SUMMARY:
This study aims to determine the efficacy of nebulising 3% hypertonic saline in improving clinical symptoms and reducing the length of hospital stay in infants with acute bronchiolitis.

DETAILED DESCRIPTION:
Bronchiolitis is the most prevalent disease in infants, especially children younger than two years old. Clinical manifestations vary from mild to severe, even life-threatening respiratory failure. Airway oedema and mucus plugging are the principal pathological features in infants with acute bronchiolitis. Nebulising 3% hypertonic saline solution may reduce these pathological changes, but the evidence remains equivocal.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients diagnosed with acute bronchiolitis from 1 to 24 months old at Can Tho Children's Hospital.

Exclusion Criteria:

* Family members do not agree to let the child participate in the study.
* Severe respiratory failure required mechanical ventilation.
* The patient left on his own during treatment.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Improve clinical severity score after three days of treatment with nebulized 3% hypertonic saline. | three days
  The clinical severity score is a validated, self-reported instrument assessing clinical severity over treatment. Possible scores range from 0 (mild) to 12 (severity).

SECONDARY OUTCOMES:
Shorten the mean length of hospital stays in infants with bronchiolitis after treatment with nebulized 3% hypertonic saline. | From admission to discharge, up to 14 days
  The mean length of hospital stays is the days from admission to discharge of all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Van VuTuong Le, MD, Principal Investigator — Can Tho University of Medicine and Pharmacy
Locations (1):
- Can Tho Children's Hospital, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication